CLINICAL TRIAL: NCT01022671
Title: Single-Arm, Open-label, Multicenter, Phase 2 Clinical Trial to Assess the Efficacy and Safety of Single-Agent Camtobell Inj.(Belotecan) Administered on A Weekly Schedule in Locally Advanced or Metastatic Non-small Cell Lung Cancer Patients Previously Treated With Chemotherapy
Brief Title: Study of Camtobell Inj (Belotecan) on Weekly Schedule in Non-small Cell Lung Cancer (NSCLC) Patients Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Asan Medical Center (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Ulsan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11NSCLC08K
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Belotecan; Camtobell inj; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — belotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belotecan (Experimental): Single arm
  Interventions: Drug: Belotecan

INTERVENTIONS:
Drug: Belotecan — 3.0 mg/m2, Day 1, 8, 15 every 4 weeks
  Other Names: Camtobell inj.

SUMMARY:
A phase II study is conducted to determine the efficacy and safety of a single agent Camtobell inj.(belotecan) on a weekly schedule in locally advanced or metastatic non-small cell lung cancer patients previously treated with chemotherapy. The usefulness of the this regimen is evaluated by response rate, median survival time, progression free survival and duration of response.

ELIGIBILITY:
Inclusion Criteria:

* 19 Years and older
* Histologically or cytologically confirmed locally advanced or metastatic NSCLC(Stage IIIB or IV)
* ≥ one measureable or evaluable lesion, <25% of the bone marrow had been irradiated
* prior platinum based chemotherapy
* ECOG PS ≤ 2
* Life expectancy > 3 months
* Adequate organ function:

  * hematology: ANC ≥ 1.5×109/L, Platelet ≥ 100×109/L, hemoglobin ≥ 9.0g/dL
  * hepatic: total bilirubin ≤ 1.5×ULN, AST/ALT ≤ 2.0×ULN, ALP ≤2.0×ULN
  * renal: serum creatinine ≤ 1.5×ULN
* Signed a written informed consent

Exclusion Criteria:

* Active infection
* Symptomatic brain lesion
* Any other type of cancer during the previous 5 years except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix
* Severe concurrent diseases
* Prior anticancer therapy within 4 weeks before enroll
* Active pregnancy test

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | every 2 cyc

SECONDARY OUTCOMES:
Overall Survival | 6 months after Last patient out
Progression Free survival | 6 months after Last patient out
Adverse event | every visit

IPD SHARING:
Plan to Share IPD: No